Creation date: January 2019.

Phase I-II clinical study to compare the safety and efficacy of Nanodrop® versus Systane® Balance in the treatment of patients with dry eye.

Protocol Code: SOPH176-1218/I-II

Protocol Version: 2.0

## Content

| 1.0 | Abbreviations | 2 | |
|----------|-----------------------------------|----|---|
| 2.0 | Objectives of the Study | 2 | 2 |
| 3.0 | Design of Study SOPH176-1218/I-II | 2 | |
| 4.0 Samp | ole Size4 | | |
| 5.0 | Sample Size Calculation | 4 | |
| 7.0 Anal | ysis Methods | 8 | |
| 8.0 | Changes | 10 | |
| 9.0 | References | 11 | |
| 10.0 Anı | nexes | 12 | |

Version 3.0

### 1.0 Abbreviations

CI Informed Consent

CRF Electronic Case Report Form

EA Adverse events

ITT Intention-to-treat population

LLS Safety call

MAVC Best corrected visual acuity
MC Concomitant medication

OSDI Ocular Surface Disease Index

PI Research Product
PP Population by protocol

PRO-176 Nanodrop®

TRL Tear break-up time
V1 Follow-up visit 1
VB Initial visit
VF Final visit

## 2.0 Objectives of the Study

Security (Phase I):

To evaluate the safety of ophthalmic application of Nanodrop® by quantifying the incidence of unexpected Adverse Events (AEs) related to the investigational product (IP).

Efficacy (Phase II):

To demonstrate the non-inferiority of Nanodrop® compared to Systane® Balance in the treatment efficacy of patients with dry eye, using the OSDI (Ocular Surface Disease Index) test score.

## 3.0 Study Design SOPH176-1218/I-II

Phase I-II, comparative, non-inferiority, active-controlled, parallel-group, double-blind, randomized clinical trial. Safety analysis comparing the visits of the first 12 patients in the Nanodrop® group. If fewer than 20% of unexpected adverse events (AEs) related to the investigational product occur, recruitment continues until the sample for the efficacy analysis is complete.

## 3.1 Duration of treatment

30 days.

## Version 3.0

Table 1. Study schedule

| Procedures | VB | V1 | VF | LIS |
|---|---|---|---|---|
| | D 1 | D 8 | D 31 to + 1 | D 37 ± 1 |
| CI Signature | Х | | | |
| Medical record | Х | | | |
| MC Evaluation | Х | Х | Х | |
| Urine pregnancy test | Х | | Х | |
| MAVC | Х | Х | Х | |
| Ocular surface stains | Х | Х | Х | |
| Tear film break-up time with fluorescein | Х | Х | Х | |
| Ophthalmological evaluation | Х | Х | Х | |
| Eligibility criteria | Х | | | |
| EA Assessment | Х | Х | Х | Х |
| PI Assignment | Х | | | |
| Delivery of PI and start of intervention | Х | | | |
| Delivery of the PI and start of intervention | Х | | | |
| Delivery of patient materials and instructions for completion (Subject Diary) | Х | | | |
| Evaluation of the Diary of the subject | | Х | Х | |
| Adherence assessment | | Х | Х | |
| Continuity assessment of the subject | | Х | Х | |
| Return of PI and Subject's Diary | | | Х | |

CI: Informed Consent; BCVA: Best Corrected Visual Acuity; OSDI: Ocular Surface Disease Index; AE: Adverse Event; PI: Investigational Product; MC: Concomitant Medication.

#### 4.0 Sample Size

An estimated 63 subjects (both eyes) per treatment arm are planned (Phase I: 12 subjects / Phase II: 114 subjects).



Figure 1. Suggested workflow. ITT: Intention-to-treat population; PP: Per-protocol population.

#### 5.0 Sample Size Calculation

For the sample size calculation, changes in the OSDI (Ocular Surface Dehydration Index) questionnaire score were considered, in studies with ocular lubricants in patients with dry eye disease (DED), as the primary efficacy variable.

PRO-176 (Nanodrop®; Laboratorios Sophia, SA de CV) is expected to be non-inferior to its comparator (Systane® Balance; Alcon Research Ltd, Fort Worth, TX, USA), according to the following working hypotheses:

$$H_0: \varepsilon \leq \delta$$

$$H_1: \varepsilon > \delta$$

Where  $\mu_A - \mu_B = \epsilon$  is the true difference in means between the test treatment (PRO-176) and the active control (Systane® Balance). Where  $\delta$  is the non-inferiority margin, and the ratio of the sample sizes between the two groups is given by:

$$k = \frac{n_A}{n_B}$$

Calculations were performed using the non-inferiority equation for two means and for statistical power (Chow et al., 2008).

$$n_A = k n_B \ y \ n_B = \left(1 + \frac{1}{k}\right) \left(\sigma \frac{z_{1-\alpha} + z_{1-\beta}}{\mu_A - \mu_B - \delta}\right)^2$$

$$1-\beta=\theta(z-z_{1-\alpha})+\theta(-z-z_{1-\alpha}) \ , \ z=\frac{\pi_A-\pi_B-\delta}{\sigma\sqrt{\frac{1}{n_A}+\frac{1}{n_B}}}$$

Where  $\sigma$  is the standard deviation, k=nA/nB is the agreement ratio, $\theta$  is the standard Normal distribution function,  $\alpha$  is the type I error (confidence interval),  $\beta$  is the type II error (meaning that 1- $\beta$ corresponds to the power) and  $\delta$  is the test margin.

With a power of 80% ( $\beta$ =0.20), a significance level of 0.05 ( $\alpha$ ) and a non-inferiority margin ( $\delta$ ) of -5 points on the OSDI score (Grubbs et al., 2014; Labetoulle et al., 2017; Pérez-Balbuena et al, 2016).

The calculation was based on the study by Benitez-Del-Castillo et al., 2016. Phase I and II clinical study. A total of 156 healthy subjects and patients with DED were enrolled. The Phase I study included 30 healthy volunteers; it was a single-center, parallel-group, open-label study. Phase II was a multicenter, double-blind study. In Phase I, SYL1001 was administered at 1.125% and 2.25% doses, and in Phase II, at 0.375% and 0.75%. After 10 days of treatment, the primary efficacy variable was the effect on the OSDI score. OSDI scores were significantly reduced compared to baseline (p<0.01) for all treatments in both Phase I and Phase II. No statistical differences were observed between treatments.

The sample size calculation was performed considering a reduction in the OSDI score of 17.6 points for the placebo group at their final visit versus a reduction of 16.5 points for the treated group. Considering a  $\ddot{y}$  of 17.1, a similar reduction in the OSDI score is expected for both treatments, with no statistically significant differences at their final visit.

The calculation was performed using the online tool: http://powerandsamplesize.com.

The estimated sample size was 101 subjects (51 subjects per arm), which was increased by 25% to account for potential losses (25 subjects). The estimated number of subjects (both eyes) was 126.

## 6.0 Analysis Plan

The variables to be considered in the protocol are described below.

Primary efficacy outcome variables:

· OSDI test score.

Secondary efficacy outcome variables:

- · Changes in best corrected visual acuity (BCVA).
- Changes in corneal and conjunctival staining with lissamine green.
- · Corneal and conjunctival staining changes with fluorescein.
- Changes in tear film break-up time (TRL) with fluorescein.

Security Variables

Primary Safety outcome variable:

• Incidence of unexpected adverse events (AEs) related to the drug.

## Secondary safety outcome variable:

• Incidence of expected AEs.

Table 2. Operational Definition of the Variables

| Variable | Definition | Definition | Scale of | Category |
|---|---|---|---|---|
| | Conceptual | Operational | measurement | |
| Events | Any event | The events | Nominal • Frequency | uency: |
| adverse | | adverse | | Subjects presenting AE/Total number of |
| | adverse doctor | effects manifested | | exposed subjects. |
| | that occurs in a patient | during the | | expected dubjects. |
| | or clinical research | conduct of the | | Intensity: |
| | subject who was | study will be | | 0= Mild |
| | administered a | collected | | 4- Madanata |
| | | | | 1= Moderate |
| | nharman autical aredus | through the | | 2= Severe |
| | pharmaceutical produc | electronic CRF. | | Causality: |
| | that, not necessarily | ologicino ora . | | - Causanty. |
| | has a relationship | | | 0=Probably or possibly related. |
| | causal with this | | | |
| | treatment. | | | 1=Unlikely related. |
| Ocular | The OSDI is a | The evaluator | Continue | Score: |
| Surface | questionnaire | will apply | | |
| Disease Index | designed to | the questionnaire | | |
| Score | establish a severity | to the | | OSDI |
| | and | subject and | | $= \frac{(Suma\ del\ puntaje)25}{\#\ de\ respuestas\ contestada}$ |
| | classification of the | allow him to do so | | # de respuestas contestadas |
| (OSDI). | dry eye according to | answer in | | |
| | its symptoms. | calm | | |
| | | without any kind | | |
| | | of pressure | | |
| | | and/or coercion. See | | |
| | | Annex 1. OSDI. | | |
| Changes in | Visual acuity | Booklet of | Quantitative | Fraction, normal value = 0.6 to 2.0 |
| corrected | corrected (BCVA) is a | Snellen | discreet. | |
| visual | test of visual function. | | | |
| acuity | | | | |
| (BCVA). | Spatial VA is the ability | | | |
| | to distinguish | | | |
| | separate | | | |
| | elements of | | | |
| | an object and identify | | | |
| | them as | | | |
| | a whole. It is | | | |
| | | | | Daga 6 12 |

# Version 3.0

| | It quantifies the minimum angle of separation | | | |
|---|---|---|---|---|
| | (located at the nodal point of the | | | |
| | eye) between two objects that allows | | | |
| | them to be perceived as separate | | | |
| | objects. | | | |
| Changes of | Detection of | Observation | Qualitative | Degrees: |
| corneal | epithelial | direct with slit | Ordinal | The staining is presented in a series of panels |
| and | defects in the | lamp, Oxford | | (AE). The staining points range from 0-5 for |
| conjunctival<br>staining with green | conjunctiva and cornea. | scale | | each panel and from 0-15 for the total |
| lissamine. | comea. | graduation. | | exposed area of conjunctiva and cornea. |
| | | See Annex 2. | | |
| | | Oxford scale. | | |
| Corneal and | Detection of | Direct observation | Qualitative | Degrees: |
| | | The staining is presented in a series of panels | | |
| conjunctival | | | (AE). The staining points range from 0-5 for | |
| staining changes<br>with | conjunctiva and cornea. | filter, Oxford scale | | each panel and from 0-15 for the total |
| fluorescein. | | graduation. | | exposed area of conjunctiva and cornea. |
| | | See Annex 2. | | |
| | | Oxford scale. | | |
| Changes in | The stability of the | It will be measured at | Quantitative | Normal: > 10 seconds. |
| tear film break- | Tear film is usually | end of a blink and | continues. | |
| up time (TRPL) | evaluated | you will be asked | | |
| with | clinically by the | not to blink | | |
| fluorescein. | TRL. This involves | immediately<br>until the tear | | |
| | instilling | film on the | | |
| | fluorescein on the ocular | cornea | | |
| | surface to allow | breaks. | | |
| | visualization of the tear film and measure | | | |
| | the time it takes for the | | | |
| | tear film to break up | | | |
| | after the last blink. | | | |

#### 7.0 Methods of Analysis

Statistical analysis will be performed by staff of Laboratorios Sophia, SA de CV. The statistical program SPSS version 19.0 (IBM Corporation, Armonk, NY, USA) will be used.

The designated personnel will be blinded to the intervention groups. Coding will be performed using consecutive numbers for each intervention group.

The data will be collected and organized in an Excel spreadsheet (Microsoft®

Office). The data will then be exported to the SPSS software platform. The variables will be categorized according to their nature (see Table 2).

Study participants will be identified by a number and their initials.

The initials of the subject of study will be obtained starting with the first letter of the name, followed by the first letter of the first surname and the first letter of the second surname, obtaining a maximum of three letters. In case the person has two names or a compound surname, the first letter will always be used.

#### Example:

To. Arieh Daniel Mercado Carrizalez B. Juan De la Torre Orozco

to. Initials: AMC b. Initials: JDO

Once the subject has been selected, they will be assigned a number that will identify them throughout the study. This code will consist of eight numbers in the following order from left to right:

• Three digits of the molecule under study according to the sponsor's designation. • Two digits corresponding to the research center number. • Three digits of the consecutive number assigned to its inclusion at the research center.

Subjects will be divided into two equal groups, which will be randomly and blindly assigned to one of the PI, PRO-176 or Systane® Balance (assignment (1:1). Which will be administered based on the dosage described in the protocol.

A preliminary safety analysis will be performed upon completion of follow-up of subject 12 in the Nanodrop® group (Phase I).

If fewer than 20% of unexpected drug-related AEs occur in the Nanodrop® group, enrollment for the efficacy analysis (Phase II) will be completed. Otherwise, the study will be terminated.

The results of the continuous quantitative variables will be presented in measures of central tendency: mean, standard deviation and ranges, see table 2.

The Kolmogorov-Smirnov and Shapiro Wilk test will be performed to determine whether the distribution is normal in the results obtained in each study group (Haffajee et al., 1983).

Version 3.0

The statistical analysis of continuous **quantitative variables** to find significant differences (p) will be as follows:

- Intra-group analysis: will be determined using the Wilcoxon rank test, for quantitative variables (Woolson, 2008).
- Between-group analysis: differences between groups will be analyzed using the Student t-test or the Mann-Whitney U statistic if applicable (it will be used to test whether a group of data comes from the same population).

The level of difference to consider significance will be an alpha (ÿ) of 0.05 or less. It will be considered a 95% CI for non-inferiority criteria (Schumi & Wittes, 2011; Easty et al., 2006).

The result of the nominal and ordinal qualitative variables will be presented in frequencies, proportions and percentages, see table 2.

Statistical analysis to identify significant differences in **qualitative variables** will be performed by creating 2x2 contingency tables and will be carried out as follows:

- Intra-group difference: McNemar's test (Klingenberg & Agresti, 2006). This test is applied to 2x2
  contingency tables with a dichotomous trait, with matched subject pairs, to determine whether
  the marginal frequencies of the row and column are equal (marginal homogeneity).
- Difference between groups: Chi-square test (X 2) Pearson's or Fisher's exact test in values expected under 5.

The level of difference to consider significance will be an alpha (ÿ) of 0.05 or less.

For the reporting of adverse events, all eyes of participants who were randomized to an intervention group after the baseline visit will be considered.

The final results report will be displayed in tables or graphs, as appropriate.

Subjects who meet a minimum adherence of 70% will be included in the statistical analysis to meet the study objective, based on the weight of the PI. In cases where the container is not returned or has not been physically intact, adherence will be measured using the subject's diary.

## Version 3.0

The investigational drug will be considered safe and effective when there are no clinical and statistical differences in all primary outcome variables, with respect to its comparator.

(Systaine® Balance).

Table 3. Triangulation of concepts

| Variable Type Varia | able A | A1 B1 B2 C1 C2 D1 E1 E2 E3 | | | |
|---|---|---|---|---|---|
| Background | | | | | |
| A1 | Demographics | OT | | | |
| Basal | | | | | |
| B1 | Medical record | DΤ | | | |
| B2 | Comprehensive ophthalmological evaluation | DT | ТВ ТВ | ТВ | |
| Security | | | | | |
| C1 | Unexpected/related AEs | ТВ | ТВ | ТВ ТВ ТВ | |
| C2 | EAs | ТВ | ТВ | ТВ ТВ ТВ | |
| Effectiveness | | | | | |
| D1 | OSDI | DB | | DB | |
| Secondary outcome | | | | | |
| E1 | MAVC | | DB TB TB | DM | |
| E2 | Ocular surface stains | | DB TB TB | DM | |
| E3 | Tear film time | | DB TB TB | | DM |
| D: Descriptive statist | ics; T: 2x2 contingency table; B: Bivariate analysis; | M: Multivari | ate analysis. | | |

## 8.0 Changes

The following numerals were changed to match the current version of the protocol:

- 2.0 Study objectives (Effectiveness; phase II).
- \_ 3.0 Study design.
- Table 1. Study schedule.
- 5.0 Sample size calculation.
- 7.0 Methods of analysis, referring to adhesion.

## Author of the document:

Clinical Operations.

Sophia Laboratories, SA de CV

Av. Paseo del Norte 5255, Guadalajara Technology Park.

45010, Zapopan, Jalisco, Mexico.

### 9.0 References

- Benitez-Del-Castillo JM, Moreno-Montañés J, Jiménez-Alfaro I, et al. Safety and efficacy clinical trials for SYL1001, a novel short interfering RNA for the treatment of dry eye disease. Invest Ophthalmol Vis Sci, 2016; 57:6447-6454.
- 2. Chow et al. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series, 2008: Chapter 4, page 85.
- 3. Grubbs JR, et al. A review of quality of life measures in dry eye questionnaires. Cornea, 2014; 33(2): 215-218.
- 4. Haffajee A., Socransky S. and Lindhe J. Comparison of statistical methods of analysis of data from clinical periodontal trials. *J Clin Periodontol*, 1983; 10: 247-256. 5. http://
- powerandsamplesize.com, equations based on; Chow et al. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series, 2008.
- 6. ICH E2A. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartitite Guideline. Clinical safety data management: definitions and standards for expedited reporting. October 1994.
- 7. Klingenberg B. and A. Agresti A. Multivariate extension of McNemar's test. *Biometrics*, 2006. vol. 62, pp. 921-928.
- 8. Labetoulle M, et al. Osmoprotectants, carboxymethylcellulose and hyaluronic acid multi-ingredient eye drop: a randomized controlled trial in moderate to severe dry eye. Eye, 2017; 31:1409-1416.
- Pérez-Balbuena AL, et al. Efficacy of a fixed combination of 0.09% xanthan gum/0.1% chondroitin sulfate preservative free
  vs polyethylene glycol/propylene glycol in subjects with dry eye disease: a multicenter randomized controlled trial. BMC
  Ophthalmol, 2016; 16:164.
- 10. Woolson R. Wilcoxon signed-rank test. Wiley Encuclopedia of Clinical Trials, 2008, pp. 1-3.
- 11. Schumi J and Wittes JT. Through the looking glass: understanding non-inferiority. trials, 2011; 12:106.
- 12. Easty DL, Nemeth-Wasmer G, Vounatsos JP., et al. Comparison of a non-preserved 0.1% T-Gel eye gel (single dose unit) with a preserved 0.1% T-Gel eye gel (multidose) in ocular hypertension and glaucomatous patients. Br J Ophthalmol, 2006; 90:574-578.

#### 10.0 Annexes

### 10.1 Ocular Surface Disease Index

The OSDI (ocular surface disease index) test is a simple test designed to establish the severity and classification of dry eye based on its symptoms.

Please answer the following questions by checking the box that best represents your answer:

### 1. Have you experienced any of the following changes during the last week?

| | | FREQUENCY | | | |
|---|---|---|---|---|---|
| | Throughout<br>moment | Almost in everything moment | 50% of the time | Almost in no<br>moment | In no case<br>moment. |
| Light sensitivity. | 4 | 3 | 2 | 1 | 0 |
| Gritty feeling in the eyes. | 4 | 3 | 2 | 1 | 0 |
| Eye pain | 4 | 3 | 2 | 1 | 0 |
| Blurred vision. | 4 | 3 | 2 | 1 | 0 |
| Poor vision. | 4 | 3 | 2 | 1 | 0 |
| | 1 | 1 | | Subtotal: | |

# 2. Have you had eye problems that have limited or prevented you from performing any of the following actions? during the last week?

| | | FREQUENCY | | | |
|---|---|---|---|---|---|
| | Throughout<br>moment | Almost in everything moment | 50% of the time | Almost in no<br>moment | In no case<br>moment. |
| Read. | 4 | 3 | 2 | 1 | 0 |
| Driving at night. | 4 | 3 | 2 | 1 | 0 |
| Working on a computer or using an ATM. | 4 | 3 | 2 | 1 | 0 |
| Watch television. | 4 | 3 | 2 | 1 | 0 |
| | • | | | Subtotal: | |

#### 3. Have you experienced eye discomfort in any of the following situations during the last week?

| | FREQUENCY | | | | |
|---|---|---|---|---|---|
| | Throughout<br>moment | Almost in everything moment | 50% of the time | Almost at no time | Not at any<br>time. |
| Wind. | 4 | 3 | 2 | 1 | 0 |

# SOPH176-1218/I-II

# Statistical Analysis Plan

# Version 3.0

| Low humidity (dry) places. | 4 | 3 | 2 | 1 | 0 |
|-----------------------------|---|---|---|-----------|---|
| Areas with air conditioned. | 4 | 3 | 2 | 1 | 0 |
| | | | | Subtotal: | |

## 10.2 Oxford Scale

| PANEL | Grade | Criteria |
|-------|-------|-----------------------------------------------|
| A | 0 | Equal to or less than panel A |
| В | 1 | Equal to or less than panel B, greater than A |
| С | II | Equal to or less than panel C, greater than B |
| D | III | Equal to or less than panel D, greater than C |
| E | IV | Equal to or less than panel E, greater than D |
| >E | V | Greater than panel E |